CLINICAL TRIAL: NCT05116124
Title: Inflammatory Parameters as Predictive Factors for Complicated Appendicitis
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Tâmega e Sousa (Other)
Responsible Party: Principal Investigator, Ana Ribeiro, Principal Investigator, Centro Hospitalar do Tâmega e Sousa
Other Study IDs: CHR123456
Record Dates: First submitted 2021-10-19; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - uncomplicated appendicitis
  Interventions: Other: dosing of inflammatory parameters
- Group 2 - complicated appendicitis
  Interventions: Other: dosing of inflammatory parameters

INTERVENTIONS:
Other: dosing of inflammatory parameters — View and register the dosing of inflammatory parameters

SUMMARY:
Acute appendicitis is a major cause of acute abdomen. Although its diagnosis is clinical, it is often supported by complementary diagnostic tests. Sometimes, delay in diagnosis can lead to worsening of the clinical picture, resulting in a complicated acute appendicitis. Some series have studied some clinical and analytical parameters as possible predictors of complicated acute appendicitis.

A retrospective analysis of patients admitted for acute appendicitis and undergoing appendectomy between January 2014 and December 2017 was performed in order to assess the possible existence of preoperative analytical predictive factors for complicated acute appendicitis (such as leukocytosis, C-reactive protein and ratio between neutrophils and lymphocytes).

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted for acute appendicitis

Exclusion Criteria:

* excluded if no existence of dosing of all the inflammatory parameters cited above

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for acute appendicitis
Sampling Method: Probability Sample
Enrollment: 841 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
C-reactive protein dosage | 4 years
Leukocytosis dosage | 4 years
Ratio between neutrophils and lymphocytes dosage | 4 years

IPD SHARING:
Plan to Share IPD: Undecided